CLINICAL TRIAL: NCT03331952
Title: Monitoring Pneumococcal Conjugate Vaccine Introduction in Cambodia: A Study of Streptococcus Pneumoniae Colonisation, Pneumonia and Invasive Disease in Cambodian Children
Brief Title: A Study of Streptococcus Pneumonia Colonisation and Invasive Disease in Cambodian Children
Acronym: PCV
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: COMRU1501
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Streptococcal Pneumonia
Keywords: Streptococcal Pneumonia; Pneumococcal Conjugate Vaccine
MeSH Terms: conditions — Pneumonia | interventions — Prospective Studies; Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Invasive pneumococcal disease study (PCV-D): Prospective study of children with invasive pneumococcal disease / probable bacterial meningitis (PCV-D)
  Clinical procedures
  At study enrolment:
  * Admission clinical findings / laboratory results will be recorded.
  * A questionnaire will be administered to the parent / guardian or caretaker to assess the child's immunisation status, household structure, environmental exposures, and recent antimicrobial use.
  Radiology procedures As part of routine clinical management at AHC, a digital chest radiograph (CXR) may be performed as part of a child's diagnostic work up. CXRs will be read and interpreted primarily by the AHC radiologists. All CXR will subsequently be re-read by two study clinicians and interpreted according to the WHO paediatric radiologic pneumonia criteria.
  Laboratory procedures
  • Residual routine clinical specimens further analysed as part of the study protocol:
  * Blood and cerebrospinal fluid culture specimens.
  * EDTA / serum specimens.
  * Urine.
  Interventions: Other: Prospective study
- Pneumonia study (PCV-P): Prospective study of children hospitalised with clinical and/or radiologic pneumonia (PCV-P)
  Clinical procedures As described for PCV-D.
  Radiology procedures As part of routine clinical management at AHC, a digital chest radiograph (CXR) is performed on all children with an admission diagnosis of pneumonia. CXRs will be handled as described for PCV-D.
  Laboratory procedures
  * Study specific specimens:
    o Nasopharyngeal swab at enrolment.
  * Residual routine clinical specimens further analysed as part of the study protocol:
    * As described for PCV-D.
  Interventions: Other: Prospective study
- Pneumococcal colonisation study (PCV-C): Cross-sectional pneumococcal colonisation surveys in children attending the AHC out-patient department (PCV-C)
  Three annual surveys, enrolling 450 children each year, will be done to identify and characterise pneumococcal nasopharyngeal colonisation in AHC out-patient department (OPD) attendees.
  Clinical procedures
  • Subjects will be recruited from the OPD waiting area after nurse triage. A questionnaire will be administered to the parent / guardian or caretaker to assess the child's immunisation status (by review of the handheld immunisation card where possible), household structure, environmental exposures, and recent antimicrobial use.
  Laboratory procedures • Study specific specimens:
  o Nasopharyngeal swab at enrolment. A nasopharyngeal swab will be collected from each participant and these will be processed as described for PCV-P.
  Interventions: Other: Cross-sectional surveys

INTERVENTIONS:
Other: Prospective study — To identify and characterise patients with culture proven invasive pneumococcal disease or probable bacterial meningitis over the first three years after PCV13 introduction in Cambodia in January 2015.
  Groups: Invasive pneumococcal disease study (PCV-D)
Other: Prospective study — To identify and characterise patients hospitalised with clinical and/or radiologic pneumonia over the first three years after PCV13 introduction in Cambodia in January 2015
  Groups: Pneumonia study (PCV-P)
Other: Cross-sectional surveys — Three annual surveys, enrolling 450 children each year, will be done to identify and characterise pneumococcal nasopharyngeal colonisation in AHC out-patient department (OPD) attendees
  Groups: Pneumococcal colonisation study (PCV-C)

SUMMARY:
Streptococcus pneumoniae (the pneumococcus) remains a leading cause of childhood mortality and morbidity. Between 2007 and 2012, Angkor Hospital for Children (AHC), Siem Reap, Cambodia documented that S. pneumoniae was responsible for around 10% of bloodstream infections in hospitalised children, with a case fatality rate of 15.6%.

The use of pneumococcal conjugate vaccines (PCV), covering between 7 and 13 of the >90 pneumococcal serotypes, has resulted in significant declines in invasive pneumococcal disease (IPD) incidence in countries where they are included in routine childhood immunisation schedules. Paediatric radiologic pneumonia incidence is also reduced by PCV, but the impact on clinical pneumonia is minimal. The vaccines have had an effect on reducing the burden of drug resistant IPD, although this may not be sustained. Given the large number of serotypes not included in the current PCV formulations, it is not surprising that initial declines in overall IPD incidence have been eroded by, for the time being, small increases in IPD due to non-vaccine serotypes. To date most data on this serotype replacement disease has come from high-income countries. It less clear how much serotype replacement will occur in low and middle income countries, where pre-PCV disease incidence is generally higher and other factors, such as unregulated antimicrobial consumption, may play a role in encouraging non-vaccine serotype infections.

Nasopharyngeal colonisation by S. pneumoniae is common in childhood and is an essential prerequisite for invasive disease. Surveillance of pneumococcal colonisation can provide important data regarding serotype replacement and disease-associated serotypes, and may also allow prediction of likely IPD incidence changes post-vaccine introduction. A recent study of pneumococcal colonisation in children attending the AHC out-patients has documented an overall colonisation prevalence of approximately 65%.

In January 2015, Cambodia will introduce the 13-valent PCV (PCV13; serotypes covered 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19F, 19A, 23F). The vaccine will be rolled out nationally with a 3+0 dosing schedule (6, 10 and 14 weeks) and no catch up campaign. There is no robust national surveillance system in place to monitor the effects of PCV13 introduction.

ELIGIBILITY:
Group1: PCV-D

Inclusion:

* Age: 0 - 59 months on the day of assessment / culture AND
* S.pneumoniae identified from a normally sterile site culture. OR
* WHO Coordinated Invasive Bacterial Vaccine Preventable Diseases (IB-VPD) Surveillance Network Case Definition for probable bacterial meningitis. Clinically suspected meningitis and a CSF examination with at least one of:

  * Turbid appearance.
  * Leucocytosis (WBC count of >100 cells/mm3).
  * Leucocytosis (10-100 cells/mm3) AND either an elevated protein (>100 mg/dL) or decreased glucose (<2.2 mmol/L).

Exclusion:

* Previous enrolment within the last 14 days.
* Parent / guardian or caretaker refused consent.

Group2: PCV-P

Inclusion:

* Age: 0 - 59 months on the day of admission AND
* Admission to the IPD, ER/ICU, or NICU/SCBU. AND
* Meets the WHO Coordinated Invasive Bacterial Vaccine Preventable Diseases (IB-VBD) Surveillance Network pneumonia / severe pneumonia case definition:

  * Cough and/or difficulty breathing. AND
  * Tachypnoea OR
  * Inability to breast feed or drink.
  * Vomiting everything.
  * Convulsions.
  * Prostration/lethargy.
  * Chest indrawing.
  * Stridor when calm.

Exclusion:

* Previous enrolment within the last 14 days.
* Parent / guardian or caretaker refused consent.

Group3: PCV-C

Inclusion:

• Age: 0 - 59 months on the day of recruitment

Exclusion:

* Parent / guardian or caretaker reports symptoms of potential acute lower respiratory tract illness.
* Triage nurse selects child for doctor review / hospital admission.
* Previous enrolment in the current annual survey.
* Parent / guardian or caretaker refused consent.

Ages: 0 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Group1: This is a prospective study to identify and characterise patients with culture proven invasive pneumococcal disease or probable bacterial meningitis over the first three years after PCV13 introduction in Cambodia in January 2015.
  Group2: This is a prospective study to identify and characterise patients hospitalised with clinical and/or radiologic pneumonia over the first three years after PCV13 introduction in Cambodia in January 2015.
  Group3: Three annual surveys, enrolling 450 children each year, will be done to identify and characterise pneumococcal nasopharyngeal colonisation in AHC out-patient department (OPD) attendees.
Sampling Method: Non-Probability Sample
Enrollment: 4111 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Invasive pneumococcal disease hospitalisation rates | 3 years
Characteristics of invasive S. pneumoniae isolates in children <5 years of age admitted to Angkor Hospital for Children, in relation to national introduction of PCV13 in Cambodia | 3 years

SECONDARY OUTCOMES:
Changes in pneumonia (both clinical and radiologic) hospitalisation rates in children <5 years of age, in relation to national introduction of PCV13 in Cambodia | 3 years
Pneumococcal colonisation prevalence | 3 years
Antimicrobial susceptibility profiles in relation to national introduction of PCV13 | 3 years
Serotype in relation to national introduction of PCV13 | 3 years
Genotype in relation to national introduction of PCV13 | 3 years
Compare pneumococcal serotype colonisation in pneumonia cases with children attending the hospital out-patients for minor illnesses | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Angkor Hospital for Children, Siem Reap, Cambodia